CLINICAL TRIAL: NCT03097991
Title: Randomized Controlled Trial of Prenatal Coparenting Intervention for African American Fragile Families
Brief Title: Randomized Controlled Trial of Prenatal Coparenting Intervention (CoparentRCT)
Acronym: CoparentRCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of South Florida (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: NIH 5R01HD082211-01; R01HD082211 (NIH)
Record Dates: First submitted 2016-12-02; First posted 2017-03-31 (Actual); Results first posted 2022-12-15 (Actual); Last update posted 2022-12-15 (Actual); Status verified 2022-01

CONDITIONS: Parenting
Keywords: Coparenting Unmarried African-American Prenatal

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention: Treatment as Usual + Focused Coparenting Consult (Experimental): Receipt of Treatment As Usual/Resource and Referral supports, plus opportunity to complete six 90-minute Focused Coparenting Consultation (FCC) sessions followed by one postnatal booster session designed to strengthen the mother-father coparenting alliance
  Interventions: Behavioral: Focused Coparenting Consultation
- Control: Treatment as Usual (No Intervention): Receipt of TAU/Resource and Referral supports

INTERVENTIONS:
Behavioral: Focused Coparenting Consultation — Six 90-minute sessions completed within 10 weeks address importance of coparenting for child development; overcoming challenges to coparenting collaboratively; anger and conflict management and communication skills. Parents develop a coparenting plan to support one another's involvement as parents to the baby. A 90-minute booster session one month after the baby's birth reinforces lessons learned in the 6-session intervention.
  Arms: Intervention: Treatment as Usual + Focused Coparenting Consult

SUMMARY:
This R01 tests through RCT methodology efficacy of a new intervention designed specifically to aid development of positive coparenting alliances between at-risk (unmarried, uncoupled, low income) African American mothers and fathers having a first baby together.

DETAILED DESCRIPTION:
Seventy-five randomly-assigned control group families will receive county services as-usual (TAU) for pregnant parents and assistance of the partnering health and human service agencies with referrals to desired services, while 75 experimental group families will receive the same services and aid, plus a 6-session prenatal intervention with a post-natal booster session. The intervention addresses the importance of safe, healthy families for early infant development, the impact a cooperative and sustained coparenting alliance can have in promoting positive infant development, challenges unmarried parents face cultivating a coparenting alliance together when their commitment to one another as romantic or married partners is in doubt, and ways to surmount these obstacles, maintain rapport, and sustain a strong alliance. Participating families, both at intake (prior to the intervention) and then again at 3 and 12 months post-partum, will report beliefs about fatherhood; extent of depressive symptomatology; and quality of the mother-father partnership, including intimate partner violence (IPV). State-of-the-field coparenting observations will be conducted at each follow-up, along with new measures of perceived coparenting communication and respect, father engagement, parent stress, and (at 12 months) infant socioemotional adjustment. Analyses will examine impact of the intervention on promoting more supportive, coordinated post-partum coparenting alliances and more positive adult and infant outcomes. Exploratory analyses will examine questions relevant to father associations with child adjustment and whether the dyadic coparent intervention has an impact on IPV.

ELIGIBILITY:
Inclusion Criteria:

An applicant is considered eligible if the pregnancy is the mother's first with the baby's father; the mother and father are unmarried; and reported income places at or below the county and state poverty line. The target population is African American, but mixed race parents may also enroll so long as at least one parent is African American. Minor parents will be recruited only if legally emancipated or with consent of their parent or guardian (with an exception allowed if minor parent is estranged from parent or LAR). If a potential participant reports a prior history of IPV, s/he may still be eligible for participation pending a more detailed assessment completed by trained project staff using the Danger Assessment Scale (Campbell, 2003).

Exclusion Criteria:

Families are excluded if either partner 1) has recently (within the past year) been arrested and convicted for violence (assault) perpetrated against someone other than a current or former partner who is the co-parent of one of their children; 2) demonstrates evidence of psychotic symptoms or suicidal ideation on the Brief Symptom Inventory; or 3) is deemed high risk or in need of more intensive intervention. Risk determination is made by weighing the parent's report on the Danger Assessment Scale (DAS). As a rule of thumb, DAS scores of 9 or higher result in automatic exclusion from the study. However, even with a score below 9, a parent may disclose one or more of the following issues during administration of the DAS - any of which would result in exclusion from the study: 1) parent reports requiring medical care because of significant injuries due to partner's violence, 2) parent says she fears for her life, 3) parent reports that the partner has threatened with a weapon and owns a gun or has a gun in the household; 4) parent reports that the partner has threatened to kill her; 5) parent reports that violence has escalated recently; 6) parent reports the partner's use of illicit drugs such as cocaine, methamphetamines, hallucinogens, or opiates.

Ages: 14 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 276 (Actual)
Dates: Start 2015-09-26 (Actual); Primary Completion 2021-12-18 (Actual); Study Completion 2021-12-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James P McHale, PhD, Principal Investigator — University of South Florida
Locations (1):
- University of South Florida, Tampa, Florida, United States

IPD SHARING:
Plan to Share IPD: Yes
Once all data collection for this project has been completed and study results published, study data stripped of all subject identifiers will be available upon request, provided through electronic means in the original data management files, to qualified researchers.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Starting 6 months after publication for 5 years.
Access Criteria: Any request for study data which meets reasonable standards of scientific integrity will be considered by the study investigators, with the expectation that any costs incurred in providing such data accrued from this project will be covered by the requesting investigator.

REFERENCES:
- [Result] McHale JP, Stover CS, Dube C, Sirotkin YS, Lewis S, McKay K. A culturally grounded prenatal coparenting intervention: Results of a randomized controlled trial with unmarried Black parents. J Fam Psychol. 2022 Jun;36(4):479-489. doi: 10.1037/fam0000965. Epub 2022 Jan 27. PMID 35084880

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: dyads (mother+father)
Period: Overall Study
Arm/Group | Intervention: Treatment as Usual + Focused Coparenting Consult | Control: Treatment as Usual
Started | 140; 70 dyads (mother+father) | 136; 68 dyads (mother+father)
3 Months Post | 88; 44 dyads (mother+father) | 102; 54 dyads (mother+father)
Completed (12 months post) | 90; 45 dyads (mother+father) | 86; 43 dyads (mother+father)
Not Completed | 50; 25 dyads (mother+father) | 50; 25 dyads (mother+father)
Not completed — Didn't meet study criteria | 8 | 0
Not completed — Withdrawal by Subject | 12 | 6
Not completed — Death of Baby | 3 | 1
Not completed — Lost to Follow-up | 24 | 38
Not completed — Adverse Event | 3 | 5

BASELINE CHARACTERISTICS:
Population: The study included two main arms/groups - Intervention (Treatment as usual +Focused Coparenting Consult) and Control (treatment as usual). The main unit of analysis was the family consisting of father and mother. However for some self-report measures, the analyses included separate comparisons between the men/women in both groups. Since for some of the analyses the unit of analysis was the dyad, the men/women arms were combined.
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention: Treatment as Usual + Focused Coparenting Consult | Control: Treatment as Usual | Total
Number analyzed (Participants) | 140 | 136 | 276
Age, Continuous [Mean (Standard Deviation); unit: years] | 25.00 (6.61) | 25.62 (7.05) | 25.31 (6.83)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 70 | 68 | 138
  Male | 70 | 68 | 138
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 0 | 6
  Not Hispanic or Latino | 134 | 136 | 270
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 123 | 117 | 240
  White | 14 | 16 | 30
  More than one race | 3 | 3 | 6
  Unknown or Not Reported | 0 | 0 | 0
History of Interpersonal Partner Violence (IPV) [Count of Participants; unit: Participants] — Self-report on instances of interpersonal partner violence within the last 12 months.
  Participants | 70 | 86 | 156

OUTCOME MEASURES:

1. Primary Outcome: System for Coding Interactions in Dyads (SCID) Positive Communication Patterns
Description: Composite of SCID observational measures of positive mother-father interaction (Problem Solving Communication**, Support**, Cohesiveness*, Withdrawal**, Positive Affect**) * Couple variable, there is only one score for the couple.
  ** Individual variable, there are two separate scores for mothers and fathers separately.
  Each sub-scale scores range from 1 to 5. Total scale scores were combined by averaging the individual and couple scales, with higher scores indicating more positive patterns in couple interaction (total scale score range 1-5).
  Change from Prenatal to 3 months post-partum is evaluated.
Time Frame: Prenatal and 3 months post-partum
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: dyads
Arm/Group | Intervention: Treatment as Usual + Focused Coparenting Consult | Control: Treatment as Usual
Number analyzed (Participants) | 74 | 88
Number analyzed (dyads) | 37 | 44
score on a scale
  Prenatal | 2.46 (0.76) | 2.53 (0.68)
  3 months | 2.25 (0.45) | 2.15 (0.56)
Statistical Analysis 1: Comparison: Intervention: Treatment as Usual + Focused Coparenting Consult vs Control: Treatment as Usual; Test type: Superiority; p = .32, Mixed Models Analysis; Slope = 1.86, Standard Error of Mean 1.86 — Group x Timepoint Effect
Statistical Analysis 2: Comparison: Intervention: Treatment as Usual + Focused Coparenting Consult vs Control: Treatment as Usual; Test type: Superiority; p = .53, Mixed Models Analysis; Slope = -.84, Standard Error of Mean 1.33 — Group Effect

2. Primary Outcome: System for Coding Interactions in Dyads (SCID) Negative Communication Patterns
Description: Composite of SCID observational measures of negative mother-father interaction (Negative Escalation*, Verbal Aggression**, Attempts to Control**, Negativity/conflict**, Coerciveness**, Dysphoric Affect**) * Couple variable, there is only one score for the couple.
  ** Individual variable, there are two separate scores for mothers and fathers separately.
  Each sub-scale scores range from 1 to 5. Total scale scores were combined by summing up the individual scales, with higher scores indicating more negative patterns in couple interaction.
  Each sub-scale scores range from 1 to 5. Total scale scores were combined by averaging the individual and couple scales, with higher scores indicating more positive patterns in couple interaction (total scale score range 1-5).
  Change from prenatal to 3 months post-partum is evaluated.
Time Frame: Prenatal and 3 months post-partum
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: dyads
Arm/Group | Intervention: Treatment as Usual + Focused Coparenting Consult | Control: Treatment as Usual
Number analyzed (Participants) | 74 | 88
Number analyzed (dyads) | 37 | 44
score on a scale
  Prenatal | 1.80 (0.67) | 1.85 (0.73)
  3 months | 1.60 (0.64) | 2.00 (0.69)
Statistical Analysis 1: Comparison: Intervention: Treatment as Usual + Focused Coparenting Consult vs Control: Treatment as Usual; Test type: Superiority; p = .07, Mixed Models Analysis; Slope = -3.04, Standard Error of Mean 1.63 — Group x Timepoint Effect
Statistical Analysis 2: Comparison: Intervention: Treatment as Usual + Focused Coparenting Consult vs Control: Treatment as Usual; Test type: Superiority; p = .69, Mixed Models Analysis; Slope = .54, Standard Error of Mean 1.36; Group Effect

3. Primary Outcome: System for Coding Interactions in Dyads (SCID) Positive Communication Patterns
Description: Composite of SCID observational measures of positive mother-father interaction (Problem Solving Communication**, Support**, Cohesiveness*, Withdrawal**, Positive Affect**) * Couple variable, there is only one score for the couple.
  ** Individual variable, there are two separate scores for mothers and fathers separately.
  Each sub-scale scores range from 1 to 5. Total scale scores were combined by averaging the individual and couple scales, with higher scores indicating more positive patterns in couple interaction (total scale score range 1-5).
  Change from prenatal to 12 months post-partum is evaluated.
Time Frame: Prenatal and 12 months post-partum
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: dyads
Arm/Group | Intervention: Treatment as Usual + Focused Coparenting Consult | Control: Treatment as Usual
Number analyzed (Participants) | 68 | 64
Number analyzed (dyads) | 34 | 32
score on a scale
  Prenatal | 2.46 (0.76) | 2.53 (0.68)
  12 months | 2.05 (0.66) | 1.99 (0.38)
Statistical Analysis 1: Comparison: Intervention: Treatment as Usual + Focused Coparenting Consult vs Control: Treatment as Usual; Test type: Superiority; p = .22, Mixed Models Analysis; Slope = 2.44, Standard Error of Mean 2.00 — Group x Timepoint Effect
Statistical Analysis 2: Comparison: Intervention: Treatment as Usual + Focused Coparenting Consult vs Control: Treatment as Usual; Test type: Superiority; p = .53, Mixed Models Analysis; Slope = .84, Standard Error of Mean 1.33 — Group effect

4. Primary Outcome: System for Coding Interactions in Dyads (SCID) Negative Communication Patterns
Description: Composite of SCID observational measures of negative mother-father interaction (Negative Escalation*, Verbal Aggression**, Attempts to Control**, Negativity/conflict**, Coerciveness**, Dysphoric Affect**) * Couple variable, there is only one score for the couple.
  ** Individual variable, there are two separate scores for mothers and fathers separately.
  Each sub-scale scores range from 1 to 5. Total scale scores were combined by averaging the individual and couple scales, with higher scores indicating more positive patterns in couple interaction (total scale score range 1-5).
  Change from prenatal to 12 months post-partum is evaluated.
Time Frame: Prenatal and 12 months post-partum
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: dyads
Arm/Group | Intervention: Treatment as Usual + Focused Coparenting Consult | Control: Treatment as Usual
Number analyzed (Participants) | 68 | 64
Number analyzed (dyads) | 34 | 32
score on a scale
  Prenatal | 1.80 (0.67) | 1.85 (0.73)
  12 months | 1.78 (0.61) | 1.91 (0.67)
Statistical Analysis 1: Comparison: Intervention: Treatment as Usual + Focused Coparenting Consult vs Control: Treatment as Usual; Test type: Superiority; p = .33, Mixed Models Analysis; Slope = -1.73, Standard Error of Mean 1.76 — Group x Timepoint Effect
Statistical Analysis 2: Comparison: Intervention: Treatment as Usual + Focused Coparenting Consult vs Control: Treatment as Usual; Test type: Superiority; p = .69, Mixed Models Analysis; Slope = .54, Standard Error of Mean 1.36 — Group Effect

5. Primary Outcome: Coparenting and Family Rating Scale (CFRS) Coparent Solidarity/Family Harmony
Description: Composite of CFRS observational measures of warmth (range 1-7), cooperation (range 1-7), and sensitivity (range 1-7) and negatively loaded disengagement (range 1-7). Total scale scores were combined by averaging up the sub-scale scores, with higher values indicating better coparent solidarity/family harmony (total scale score range 1-7).
Time Frame: 3 months post-partum
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: dyads
Arm/Group | Intervention: Treatment as Usual + Focused Coparenting Consult | Control: Treatment as Usual
Number analyzed (Participants) | 72 | 92
Number analyzed (dyads) | 36 | 46
score on a scale | 1.55 (0.60) | 1.50 (0.56)
Statistical Analysis 1: Comparison: Intervention: Treatment as Usual + Focused Coparenting Consult vs Control: Treatment as Usual; Test type: Superiority; p = .81, Mixed Models Analysis; Slope = .04, Standard Error of Mean .17 — Group Effect
Statistical Analysis 2: Comparison: Intervention: Treatment as Usual + Focused Coparenting Consult vs Control: Treatment as Usual; Test type: Superiority; p = .56, Mixed Models Analysis; Slope = .01, Standard Error of Mean .02 — Group x Timepoint Effect

6. Primary Outcome: Coparenting and Family Rating Scale (CFRS) Coparent Negativity/Hostility & Competitiveness
Description: Composite CFRS observational measures of competition (range 1-7), over stimulation (range 1-7), and verbal sparring (range 1-5).
  Total scale scores were combined by averaging up the sub-scale scores, with higher values indicating better coparent solidarity/family harmony (total scale score range 1-7).
Time Frame: 3 months post-partum
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: dyads
Arm/Group | Intervention: Treatment as Usual + Focused Coparenting Consult | Control: Treatment as Usual
Number analyzed (Participants) | 72 | 92
Number analyzed (dyads) | 36 | 46
score on a scale | 0.97 (0.49) | 0.94 (0.45)
Statistical Analysis 1: Comparison: Intervention: Treatment as Usual + Focused Coparenting Consult vs Control: Treatment as Usual; Test type: Superiority; p = .77, Mixed Models Analysis; Slope = .04, Standard Error of Mean .13 — Group Effect
Statistical Analysis 2: Comparison: Intervention: Treatment as Usual + Focused Coparenting Consult vs Control: Treatment as Usual; Test type: Superiority; p = .85, Mixed Models Analysis; Slope = -.003, Standard Error of Mean .02 — Group x Timepoint Effect

7. Primary Outcome: Coparenting and Family Rating Scale (CFRS) Coparent Solidarity/Family Harmony
Description: as for outcome 5
Time Frame: 12 months post-partum
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: dyads
Arm/Group | Intervention: Treatment as Usual + Focused Coparenting Consult | Control: Treatment as Usual
Number analyzed (Participants) | 72 | 68
Number analyzed (dyads) | 36 | 34
score on a scale | 1.49 (0.67) | 1.32 (0.62)
Statistical Analysis 1: Comparison: Intervention: Treatment as Usual + Focused Coparenting Consult vs Control: Treatment as Usual; Test type: Superiority; p = .56, Mixed Models Analysis; Slope = .01, Standard Error of Mean .02 — Group x Timepoint Effect
Statistical Analysis 2: Comparison: Intervention: Treatment as Usual + Focused Coparenting Consult vs Control: Treatment as Usual; Test type: Superiority; p = .81, Mixed Models Analysis; Slope = .04, Standard Error of Mean .17 — Group Effect

8. Primary Outcome: Coparenting and Family Rating Scale (CFRS) Coparent Negativity/Hostility & Competitiveness
Description: as for outcome 6
Time Frame: 12 months post-partum
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: dyads
Arm/Group | Intervention: Treatment as Usual + Focused Coparenting Consult | Control: Treatment as Usual
Number analyzed (Participants) | 72 | 68
Number analyzed (dyads) | 36 | 34
score on a scale | 0.90 (0.30) | 0.90 (0.46)
Statistical Analysis 1: Comparison: Intervention: Treatment as Usual + Focused Coparenting Consult vs Control: Treatment as Usual; Test type: Superiority; p = .85, Mixed Models Analysis; Slope = -.003, Standard Error of Mean .02 — Group x Timepoint effect
Statistical Analysis 2: Comparison: Intervention: Treatment as Usual + Focused Coparenting Consult vs Control: Treatment as Usual; Test type: Superiority; p = .77, Mixed Models Analysis; Slope = .04, Standard Error of Mean .13 — Group Effect

9. Primary Outcome: Perceived Coparenting Solidarity as Measured by Parenting Alliance Measure (PAM) Communication Subscale
Description: Scores on Parenting Alliance Measure range from 20 to 100 with higher scores indicating more positive perceived alliance between parents. Scores on the Communication subscale range from 17 to 85.
Time Frame: 12 months post-partum compared to 3 months post-partum
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Intervention: Treatment as Usual + Focused Coparenting Consult Women; Intervention: Treatment as Usual + Focused Coparenting Consult Men: Receipt of Treatment As Usual/Resource and Referral supports, plus opportunity to complete six 90-minute Focused Coparenting Consultation (FCC) sessions followed by one postnatal booster session designed to strengthen the mother-father coparenting alliance
  Focused Coparenting Consultation: Six 90-minute sessions completed within 10 weeks address importance of coparenting for child development; overcoming challenges to coparenting collaboratively; anger and conflict management and communication skills. Parents develop a coparenting plan to support one another's involvement as parents to the baby. A 90-minute booster session one month after the baby's birth reinforces lessons learned in the 6-session intervention.
- Control: Treatment as Usual Women; Control: Treatment as Usual Men: Receipt of TAU/Resource and Referral supports
Arm/Group | Intervention: Treatment as Usual + Focused Coparenting Consult Women | Intervention: Treatment as Usual + Focused Coparenting Consult Men | Control: Treatment as Usual Women | Control: Treatment as Usual Men
Number analyzed (Participants) | 42 | 40 | 54 | 48
score on a scale
  12 months | 71.58 (14.43) | 72.79 (14.43) | 68.81 (15.42) | 72.50 (15.44)
  3 months | 64.78 (27.9) | 65.52 (29.1) | 53.41 (31.04) | 53.43 (35.59)
Statistical Analysis 1: Comparison: Intervention: Treatment as Usual + Focused Coparenting Consult Women vs Intervention: Treatment as Usual + Focused Coparenting Consult Men vs Control: Treatment as Usual Women vs Control: Treatment as Usual Men; Test type: Superiority; p < .001, Mixed Models Analysis; Slope = 21.01, Standard Error of Mean 5.91 — Group x Timepoint
Statistical Analysis 2: Comparison: Intervention: Treatment as Usual + Focused Coparenting Consult Women vs Intervention: Treatment as Usual + Focused Coparenting Consult Men vs Control: Treatment as Usual Women vs Control: Treatment as Usual Men; Test type: Superiority; p < .001, Mixed Models Analysis; Slope = 2.98, Standard Error of Mean 4.75 — Group

10. Primary Outcome: Perceived Coparenting Solidarity as Measured by Parenting Alliance Measure (PAM) Respect Subscale
Description: Scores on Parenting Alliance Measure range from 20 to 100 with higher scores indicating more positive perceived alliance between parents. Scores on the Respect subscale range from 3 to 15.
Time Frame: 12 months post-partum compared to 3 months post-partum
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention: Treatment as Usual + Focused Coparenting Consult Women | Intervention: Treatment as Usual + Focused Coparenting Consult Men | Control: Treatment as Usual Women | Control: Treatment as Usual Men
Number analyzed (Participants) | 42 | 40 | 54 | 48
score on a scale
  12 months | 13.38 (2.28) | 13.40 (2.30) | 12.67 (2.53) | 12.85 (3.14)
  3 months | 11.67 (5.02) | 11.63 (5.24) | 10.13 (5.61) | 9.28 (6.4)
Statistical Analysis 1: Comparison: Intervention: Treatment as Usual + Focused Coparenting Consult Women vs Intervention: Treatment as Usual + Focused Coparenting Consult Men vs Control: Treatment as Usual Women vs Control: Treatment as Usual Men; Test type: Superiority; p < .05, Mixed Models Analysis; linear mixed effects; Slope = .68, Standard Error of Mean .49 — Group
Statistical Analysis 2: Comparison: Intervention: Treatment as Usual + Focused Coparenting Consult Women vs Intervention: Treatment as Usual + Focused Coparenting Consult Men vs Control: Treatment as Usual Women vs Control: Treatment as Usual Men; Test type: Superiority; p < .05, Mixed Models Analysis; Slope = .26, Standard Error of Mean .60 — Group x Timepoint

11. Primary Outcome: Intimate Partner Violence as Assessed by the Psychological Aggression Scale of the Revised-Conflict Tactics Scale (CTS2; Straus et al., 1996).
Description: Scores on the Psychological Aggression Scale range from 0 to 175 and higher scores indicate more frequent acts of psychological aggression by partner.
Time Frame: 12 months post-partum compared to 3 months post-partum
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention: Treatment as Usual + Focused Coparenting Consult Women | Intervention: Treatment as Usual + Focused Coparenting Consult Men | Control: Treatment as Usual Women | Control: Treatment as Usual Men
Number analyzed (Participants) | 42 | 35 | 54 | 43
score on a scale
  12 months | 11.91 (14.36) | 14.51 (29.06) | 20.21 (25.23) | 15.17 (26.90)
  3 months | 12.26 (20.00) | 6.91 (10.19) | 17.22 (22.32) | 15.16 (24.97)
Statistical Analysis 1: Comparison: Intervention: Treatment as Usual + Focused Coparenting Consult Women vs Intervention: Treatment as Usual + Focused Coparenting Consult Men vs Control: Treatment as Usual Women vs Control: Treatment as Usual Men; We analyzed the CTS scales "Psychological Aggression" and "Physical Assault." Inspection of the latter in the raw data and descriptives showed extremely consistent selection of the lowest value of the scale (no incidents of assault) across all respondents, so we did not conduct inferential tests; Test type: Superiority; p = .39, Mixed Models Analysis; Slope = 3.52, Standard Error of Mean 4.14 — Group
Statistical Analysis 2: Comparison: Intervention: Treatment as Usual + Focused Coparenting Consult Women vs Intervention: Treatment as Usual + Focused Coparenting Consult Men vs Control: Treatment as Usual Women vs Control: Treatment as Usual Men; Test type: Superiority; p < .005, Mixed Models Analysis; Slope = -13.38, Standard Error of Mean 4.86 — Group x Time

12. Primary Outcome: Infant Socio-emotional Competencies as Assessed by the Negative Emotionality Scale of the Infant Toddler Social Emotional Assessment (ITSEA; Carter & Briggs-Gowan, 2006)
Description: Items are rated on the following 3-point scale: (0) Not true/rarely, (1) Somewhat true/sometimes, and (2) Very true/often. A "No opportunity" code allows parents to indicate that they have not had the opportunity to observe certain behaviors (e.g., behavior with peers).
  Scores on Negative Emotionality scale which includes 13 items range from 0 to 26 with higher scores are considered indicative of a deficit or delay.
Time Frame: 12 months post-partum
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention: Treatment as Usual + Focused Coparenting Consult Women | Intervention: Treatment as Usual + Focused Coparenting Consult Men | Control: Treatment as Usual Women | Control: Treatment as Usual Men
Number analyzed (Participants) | 46 | 41 | 45 | 36
score on a scale | 6.83 (4.50) | 7.14 (3.75) | 8.73 (3.85) | 8.28 (4.56)
Statistical Analysis 1: Comparison: Intervention: Treatment as Usual + Focused Coparenting Consult Women vs Intervention: Treatment as Usual + Focused Coparenting Consult Men vs Control: Treatment as Usual Women vs Control: Treatment as Usual Men; Test type: Superiority; p = .24, Mixed Models Analysis; Slope = -1.17, Standard Error of Mean 1.25 — Group
Statistical Analysis 2: Comparison: Intervention: Treatment as Usual + Focused Coparenting Consult Women vs Intervention: Treatment as Usual + Focused Coparenting Consult Men vs Control: Treatment as Usual Women vs Control: Treatment as Usual Men; Test type: Equivalence — ANOVA found a main effect of group, F(1, 155) = 6.85, p < .05, η2G = .04; p < .05, ANOVA; Mean Difference (Final Values) = 6.85 — Group

13. Primary Outcome: Infant Socio-emotional Competencies as Assessed by the Aggression Scale of the Infant Toddler Social Emotional Assessment (ITSEA; Carter & Briggs-Gowan, 2006)
Description: Items are rated on the following 3-point scale: (0) Not true/rarely, (1) Somewhat true/sometimes, and (2) Very true/often. A "No opportunity" code allows parents to indicate that they have not had the opportunity to observe certain behaviors (e.g., behavior with peers).
  Scores on the Aggression Scale which includes 12 items range from 0 to 24 and higher scores are considered indicative of a deficit or delay.
Time Frame: 12 months post-partum
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention: Treatment as Usual + Focused Coparenting Consult Women | Intervention: Treatment as Usual + Focused Coparenting Consult Men | Control: Treatment as Usual Women | Control: Treatment as Usual Men
Number analyzed (Participants) | 45 | 41 | 43 | 36
score on a scale | 12.00 (5.09) | 18.00 (6.54) | 17.00 (6.93) | 14.00 (6.08)
Statistical Analysis 1: Comparison: Intervention: Treatment as Usual + Focused Coparenting Consult Women vs Intervention: Treatment as Usual + Focused Coparenting Consult Men vs Control: Treatment as Usual Women vs Control: Treatment as Usual Men; Test type: Superiority; p = .02, Mixed Models Analysis; Slope = -2.53, Standard Error of Mean 1.04 — Parent x Group
Statistical Analysis 2: Comparison: Intervention: Treatment as Usual + Focused Coparenting Consult Women vs Intervention: Treatment as Usual + Focused Coparenting Consult Men vs Control: Treatment as Usual Women vs Control: Treatment as Usual Men; Test type: Superiority; p = .56, Mixed Models Analysis; Slope = .45, Standard Error of Mean .78 — Group

14. Primary Outcome: Infant Socio-emotional Competencies as Assessed by the Compliance Scale of the Infant Toddler Social Emotional Assessment (ITSEA; Carter & Briggs-Gowan, 2006)
Description: Items are rated on the following 3-point scale: (0) Not true/rarely, (1) Somewhat true/sometimes, and (2) Very true/often. A "No opportunity" code allows parents to indicate that they have not had the opportunity to observe certain behaviors (e.g., behavior with peers).
  Scores on Compliance Scale which includes 8 items range from 0 to16 with lower scores considered indicative of a deficit or delay.
Time Frame: 12 months post-partum
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention: Treatment as Usual + Focused Coparenting Consult Women | Intervention: Treatment as Usual + Focused Coparenting Consult Men | Control: Treatment as Usual Women | Control: Treatment as Usual Men
Number analyzed (Participants) | 46 | 40 | 43 | 36
score on a scale | 9.00 (2.67) | 8.63 (3.09) | 8.53 (2.47) | 9.06 (3.16)
Statistical Analysis 1: Comparison: Intervention: Treatment as Usual + Focused Coparenting Consult Women vs Intervention: Treatment as Usual + Focused Coparenting Consult Men vs Control: Treatment as Usual Women vs Control: Treatment as Usual Men; Test type: Superiority; p = .30, Mixed Models Analysis; Slope = .94, Standard Error of Mean .90 — Parent x Group
Statistical Analysis 2: Comparison: Intervention: Treatment as Usual + Focused Coparenting Consult Women vs Intervention: Treatment as Usual + Focused Coparenting Consult Men vs Control: Treatment as Usual Women vs Control: Treatment as Usual Men; Test type: Superiority; p = .36, Mixed Models Analysis; Slope = -.62, Standard Error of Mean .67 — Group

15. Primary Outcome: Infant Socio-emotional Competencies as Assessed by the Sleep Scale of the Infant Toddler Social Emotional Assessment (ITSEA; Carter & Briggs-Gowan, 2006)
Description: Items are rated on the following 3-point scale: (0) Not true/rarely, (1) Somewhat true/sometimes, and (2) Very true/often. A "No opportunity" code allows parents to indicate that they have not had the opportunity to observe certain behaviors (e.g., behavior with peers).
  Scores on the Sleep Scale which includes 5 items range from 0 to 10 with higher scores considered indicative of a deficit or delay.
Time Frame: 12 months post-partum
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention: Treatment as Usual + Focused Coparenting Consult Women | Intervention: Treatment as Usual + Focused Coparenting Consult Men | Control: Treatment as Usual Women | Control: Treatment as Usual Men
Number analyzed (Participants) | 44 | 38 | 41 | 36
score on a scale | 8.00 (2.68) | 7.00 (2.92) | 9.00 (2.88) | 7.00 (2.58)
Statistical Analysis 1: Comparison: Intervention: Treatment as Usual + Focused Coparenting Consult Women vs Intervention: Treatment as Usual + Focused Coparenting Consult Men vs Control: Treatment as Usual Women vs Control: Treatment as Usual Men; Test type: Superiority; p = .17, Mixed Models Analysis; Slope = -.75, Standard Error of Mean .55 — Parent x Group
Statistical Analysis 2: Comparison: Intervention: Treatment as Usual + Focused Coparenting Consult Women vs Intervention: Treatment as Usual + Focused Coparenting Consult Men vs Control: Treatment as Usual Women vs Control: Treatment as Usual Men; Test type: Superiority; p = .48, Mixed Models Analysis; Slope = .33, Standard Error of Mean .47 — Group

16. Primary Outcome: Father Engagement as Assessed by the Activities With Child Scale (Cabrera et al., 2004).
Description: This self report consists of 34 items on which the parent reports the frequency with which the father was engaged in various activities with the child in the past month. Questions were answered on a Likert-type scale from 1 (more than once a day) to 6 (not at all); all items were reverse scored such that higher scores reflect more frequent activity.
  Father engagement is assessed across six sub-scales (Socialization - 11 items, Management- 3 items, Didactic - 7 items, Physical play/warmth - 6 items, Caregiving - 7 items) with composite scores computed by averaging responses across items.
  Scores range from 34 to 204 for the total scale. Higher scores reflect more frequent activity with the child.
Time Frame: 12 months post-partum
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention: Treatment as Usual + Focused Coparenting Consult Women | Intervention: Treatment as Usual + Focused Coparenting Consult Men | Control: Treatment as Usual Women | Control: Treatment as Usual Men
Number analyzed (Participants) | 45 | 41 | 44 | 36
score on a scale | 110.51 (44.49) | 143.61 (29.62) | 112.89 (44.81) | 136.58 (31.57)
Statistical Analysis 1: Comparison: Intervention: Treatment as Usual + Focused Coparenting Consult Women vs Intervention: Treatment as Usual + Focused Coparenting Consult Men vs Control: Treatment as Usual Women vs Control: Treatment as Usual Men; Test type: Superiority; p = .88, Mixed Models Analysis; Slope = 1.15, Standard Error of Mean 7.34 — Group
Statistical Analysis 2: Comparison: Intervention: Treatment as Usual + Focused Coparenting Consult Women vs Intervention: Treatment as Usual + Focused Coparenting Consult Men vs Control: Treatment as Usual Women vs Control: Treatment as Usual Men; Test type: Superiority; p = .38, Mixed Models Analysis; Slope = 7.94, Standard Error of Mean 9.00 — Group x Time

17. Primary Outcome: Father Involvement as Assessed by the Father Involvement Scale (Coley & Moris, 2002)
Description: A composite score based on sum of items ranges between 6 to 24 with higher scores signifying greater paternal involvement.
Time Frame: 3 months post-partum
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention: Treatment as Usual + Focused Coparenting Consult Women | Intervention: Treatment as Usual + Focused Coparenting Consult Men | Control: Treatment as Usual Women | Control: Treatment as Usual Men
Number analyzed (Participants) | 42 | 40 | 54 | 48
score on a scale | 20.21 (4.21) | 21.78 (3.01) | 18.15 (5.43) | 21.25 (3.38)
Statistical Analysis 1: Comparison: Intervention: Treatment as Usual + Focused Coparenting Consult Women vs Intervention: Treatment as Usual + Focused Coparenting Consult Men vs Control: Treatment as Usual Women vs Control: Treatment as Usual Men; Test type: Superiority; p = .07, Mixed Models Analysis; Slope = -1.89, Standard Error of Mean 1.05 — Parent x Group
Statistical Analysis 2: Comparison: Intervention: Treatment as Usual + Focused Coparenting Consult Women vs Intervention: Treatment as Usual + Focused Coparenting Consult Men vs Control: Treatment as Usual Women vs Control: Treatment as Usual Men; Test type: Superiority; p < .001, Mixed Models Analysis; Slope = 2.52, Standard Error of Mean .74 — Group

18. Secondary Outcome: Infant Eye Gaze Triangular Engagement
Description: To assess infant triangular capacities, multi-shift gaze patterns in which infant looks from one parent to another, and then rapidly redirects gaze back to the first parent after having shifted once were counted. Four categories of triangular bids were defined, which corresponded to the different affective configurations: triangular engagement (TE), triangular monitoring (TM), triangular tension (TT), and triangular protest (TP). When the affective configurations addressed to the parents were not in the same category, the one addressed to P2 was selected as determinant of the triangular bid category.
Time Frame: 12 months compared to 3 months
Population: Parents dyads with their infants were analyzed. The triad is the unit of analysis, and thus the Overall Number of Participants reflects the total of father+mother+child participants - number of triads times the three participants in each family unit.
Measure: Mean (Standard Deviation); unit: Number of looks
Units Other Than Participants: Triads
Arm/Group | Intervention: Treatment as Usual + Focused Coparenting Consult | Control: Treatment as Usual
Number analyzed (Participants) | 99 | 105
Number analyzed (Triads) | 33 | 35
Number of looks
  12 months | 2.85 (2.79) | 1.77 (2.39)
  3 months | 0.14 (0.54) | 0.17 (0.38)
Statistical Analysis 1: Comparison: Intervention: Treatment as Usual + Focused Coparenting Consult vs Control: Treatment as Usual; Test type: Superiority; p = .92, Mixed Models Analysis; Slope = -.04, Standard Error of Mean .38 — Group
Statistical Analysis 2: Comparison: Intervention: Treatment as Usual + Focused Coparenting Consult vs Control: Treatment as Usual; Test type: Superiority; p = .05, Mixed Models Analysis; Slope = 1.12, Standard Error of Mean .57 — Group x Timepoint

19. Secondary Outcome: Infant Eye Gaze Triangular Monitoring
Description: as for outcome 18
Time Frame: 12 months compared to 3 months
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: Number of looks
Units Other Than Participants: Triads
Arm/Group | Intervention: Treatment as Usual + Focused Coparenting Consult | Control: Treatment as Usual
Number analyzed (Participants) | 99 | 105
Number analyzed (Triads) | 33 | 35
Number of looks
  12 months | 1.94 (2.32) | 2.46 (3.31)
  3 months | 0.97 (1.70) | 0.85 (1.41)
Statistical Analysis 1: Comparison: Intervention: Treatment as Usual + Focused Coparenting Consult vs Control: Treatment as Usual; Test type: Superiority; p = .81, Mixed Models Analysis; Slope = .11, Standard Error of Mean .47 — Group
Statistical Analysis 2: Comparison: Intervention: Treatment as Usual + Focused Coparenting Consult vs Control: Treatment as Usual; Test type: Superiority; p = .34, Mixed Models Analysis; Slope = -.67, Standard Error of Mean .70 — Group x Timepoint

20. Secondary Outcome: Infant Eye Gaze Triangular Tension
Description: as for outcome 18
Time Frame: 12 months compared to 3 months
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: Number of looks
Units Other Than Participants: Triads
Arm/Group | Intervention: Treatment as Usual + Focused Coparenting Consult | Control: Treatment as Usual
Number analyzed (Participants) | 99 | 105
Number analyzed (Triads) | 33 | 35
Number of looks
  12 months | 1.03 (2.27) | 0.83 (1.71)
  3 months | 0.25 (0.50) | 0.34 (1.17)
Statistical Analysis 1: Comparison: Intervention: Treatment as Usual + Focused Coparenting Consult vs Control: Treatment as Usual; Test type: Superiority; p = .76, Mixed Models Analysis; Slope = -.10, Standard Error of Mean .33 — Group
Statistical Analysis 2: Comparison: Intervention: Treatment as Usual + Focused Coparenting Consult vs Control: Treatment as Usual; Test type: Superiority; p = .53, Mixed Models Analysis; Slope = .31, Standard Error of Mean .49 — Group x Timepoint

21. Secondary Outcome: Infant Eye Gaze Triangular Protest
Description: as for outcome 18
Time Frame: 12 months compared to 3 months
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: Number of looks
Units Other Than Participants: Triads
Arm/Group | Intervention: Treatment as Usual + Focused Coparenting Consult | Control: Treatment as Usual
Number analyzed (Participants) | 99 | 105
Number analyzed (Triads) | 33 | 35
Number of looks
  12 months | 0.33 (0.96) | 0.34 (0.99)
  3 months | 0.08 (0.28) | 0.11 (0.37)
Statistical Analysis 1: Comparison: Intervention: Treatment as Usual + Focused Coparenting Consult vs Control: Treatment as Usual; Test type: Superiority; p = .88, Mixed Models Analysis; Slope = -.02, Standard Error of Mean .16 — Group
Statistical Analysis 2: Comparison: Intervention: Treatment as Usual + Focused Coparenting Consult vs Control: Treatment as Usual; Test type: Superiority; p = .95, Mixed Models Analysis; Slope = .01, Standard Error of Mean .23 — Group x Timepoint

22. Other Pre Specified Outcome: Recent Depressive Symptomatology as Gauged by the Edinburgh Depression Scale (EDS; Cox et al., 1987)
Description: Scores on EDS range from 0 to 30 with higher scores indicating more depressive symptoms in the past week.
Time Frame: 3 months post-partum compared to baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention: Treatment as Usual + Focused Coparenting Consult Women | Intervention: Treatment as Usual + Focused Coparenting Consult Men | Control: Treatment as Usual Women | Control: Treatment as Usual Men
Number analyzed (Participants) | 42 | 40 | 54 | 48
score on a scale
  3 months | 4.72 (5.30) | 5.10 (4.83) | 6.15 (6.17) | 5.25 (4.89)
  Baseline | 6.69 (5.20) | 6.00 (4.89) | 7.49 (4.28) | 7.54 (5.04)
Statistical Analysis 1: Comparison: Intervention: Treatment as Usual + Focused Coparenting Consult Women vs Intervention: Treatment as Usual + Focused Coparenting Consult Men vs Control: Treatment as Usual Women vs Control: Treatment as Usual Men; Test type: Superiority; p = .47, Mixed Models Analysis; Slope = .82, Standard Error of Mean 1.13 — Group x Timepoint
Statistical Analysis 2: Comparison: Intervention: Treatment as Usual + Focused Coparenting Consult Women vs Intervention: Treatment as Usual + Focused Coparenting Consult Men vs Control: Treatment as Usual Women vs Control: Treatment as Usual Men; Test type: Superiority; p = .07, Mixed Models Analysis; Slope = -1.68, Standard Error of Mean .93 — Group

23. Other Pre Specified Outcome: Recent Depressive Symptomatology as Gauged by the Edinburgh Depression Scale (EDS; Cox et al., 1987)
Description: Scores on EDS range from 0 to 30 with higher scores indicating more depressive symptoms in the past week.
Time Frame: 12 months post-partum compared to Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention: Treatment as Usual + Focused Coparenting Consult Women | Intervention: Treatment as Usual + Focused Coparenting Consult Men | Control: Treatment as Usual Women | Control: Treatment as Usual Men
Number analyzed (Participants) | 45 | 42 | 43 | 36
score on a scale
  12 months | 5.49 (4.71) | 5.24 (5.13) | 5.40 (4.70) | 5.19 (4.60)
  Baseline | 6.69 (5.20) | 6.00 (4.89) | 7.49 (4.28) | 7.54 (5.04)
Statistical Analysis 1: Comparison: Intervention: Treatment as Usual + Focused Coparenting Consult Women vs Intervention: Treatment as Usual + Focused Coparenting Consult Men vs Control: Treatment as Usual Women vs Control: Treatment as Usual Men; Test type: Superiority; p = .68, Mixed Models Analysis; Slope = .54, Standard Error of Mean 1.32 — Group x Timepoint
Statistical Analysis 2: Comparison: Intervention: Treatment as Usual + Focused Coparenting Consult Women vs Intervention: Treatment as Usual + Focused Coparenting Consult Men vs Control: Treatment as Usual Women vs Control: Treatment as Usual Men; Test type: Superiority; p = .07, Mixed Models Analysis; Slope = -1.68, Standard Error of Mean .93 — Group

24. Other Pre Specified Outcome: Level of Individual Parenting Stress as Assessed by the Parenting Stress Index Short Form (PSI-SF; Abidin, 1995) Parental Distress Subscale
Description: Scores range from 12 to 60 on each of the three sub-scales, and total score ranges from 36 to 180; high scores on the sub-scales and PSI-SF total score indicating greater levels of stress.
Time Frame: 12 months post-partum compared to 3 months post-partum
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention: Treatment as Usual + Focused Coparenting Consult Women | Intervention: Treatment as Usual + Focused Coparenting Consult Men | Control: Treatment as Usual Women | Control: Treatment as Usual Men
Number analyzed (Participants) | 45 | 42 | 43 | 35
score on a scale
  12 months | 25.07 (8.91) | 23.24 (10.00) | 25.26 (8.23) | 25.49 (8.27)
  3 months | 26.18 (8.74) | 23.40 (9.41) | 26.04 (9.52) | 23.83 (8.18)
Statistical Analysis 1: Comparison: Intervention: Treatment as Usual + Focused Coparenting Consult Women vs Intervention: Treatment as Usual + Focused Coparenting Consult Men vs Control: Treatment as Usual Women vs Control: Treatment as Usual Men; Test type: Superiority; p = .65, Mixed Models Analysis; Slope = -.85, Standard Error of Mean 1.90 — Group
Statistical Analysis 2: Comparison: Intervention: Treatment as Usual + Focused Coparenting Consult Women vs Intervention: Treatment as Usual + Focused Coparenting Consult Men vs Control: Treatment as Usual Women vs Control: Treatment as Usual Men; Test type: Superiority; p = .50, Mixed Models Analysis; Slope = -1.65, Standard Error of Mean 2.44 — Group x Timepoint

25. Other Pre Specified Outcome: Level of Individual Parenting Stress as Assessed by the Parenting Stress Index Short Form (PSI-SF; Abidin, 1995) Difficult Child Subscale
Description: as for outcome 24
Time Frame: 12 months post-partum compared to 3 months post-partum
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention: Treatment as Usual + Focused Coparenting Consult Women | Intervention: Treatment as Usual + Focused Coparenting Consult Men | Control: Treatment as Usual Women | Control: Treatment as Usual Men
Number analyzed (Participants) | 45 | 42 | 43 | 35
score on a scale
  12 months | 21.60 (5.99) | 23.02 (6.99) | 22.26 (5.51) | 23.37 (6.45)
  3 months | 16.48 (4.36) | 18.95 (7.92) | 17.22 (5.57) | 20.40 (8.25)
Statistical Analysis 1: Comparison: Intervention: Treatment as Usual + Focused Coparenting Consult Women vs Intervention: Treatment as Usual + Focused Coparenting Consult Men vs Control: Treatment as Usual Women vs Control: Treatment as Usual Men; Test type: Superiority; p = .48, Mixed Models Analysis; Slope = .92, Standard Error of Mean 1.30 — Group
Statistical Analysis 2: Comparison: Intervention: Treatment as Usual + Focused Coparenting Consult Women vs Intervention: Treatment as Usual + Focused Coparenting Consult Men vs Control: Treatment as Usual Women vs Control: Treatment as Usual Men; Test type: Superiority; p = .27, Mixed Models Analysis; Slope = -1.92, Standard Error of Mean 1.72 — Group x Timepoint

26. Other Pre Specified Outcome: Level of Individual Parenting Stress as Assessed by the Parenting Stress Index Short Form (PSI-SF; Abidin, 1995) Parent-Child Dysfunctional Interaction Subscale
Description: as for outcome 24
Time Frame: 12 months post-partum compared to 3 months post-partum
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention: Treatment as Usual + Focused Coparenting Consult Women | Intervention: Treatment as Usual + Focused Coparenting Consult Men | Control: Treatment as Usual Women | Control: Treatment as Usual Men
Number analyzed (Participants) | 45 | 42 | 43 | 35
score on a scale
  12 months | 17.07 (5.73) | 19.51 (8.18) | 18.40 (5.55) | 19.60 (6.95)
  3 months | 20.82 (5.19) | 23.76 (7.38) | 21.06 (5.25) | 22.85 (6.28)
Statistical Analysis 1: Comparison: Intervention: Treatment as Usual + Focused Coparenting Consult Women vs Intervention: Treatment as Usual + Focused Coparenting Consult Men vs Control: Treatment as Usual Women vs Control: Treatment as Usual Men; Test type: Superiority; p = .01, Mixed Models Analysis; Slope = -1.15, Standard Error of Mean 1.22 — Group
Statistical Analysis 2: Comparison: Intervention: Treatment as Usual + Focused Coparenting Consult Women vs Intervention: Treatment as Usual + Focused Coparenting Consult Men vs Control: Treatment as Usual Women vs Control: Treatment as Usual Men; Test type: Superiority; p = .58, Mixed Models Analysis; Slope = 1.08, Standard Error of Mean 1.96 — Group x Timepoint

ADVERSE EVENTS:
Time Frame: 15 months
Description: The adverse events were collected between the date of the first subject enrollment and the date of the last study follow-up.
  This is the best estimate of the specific Time Frame and is expressed as an average duration of time for each participant.
  The adverse events reported as affecting the individual involved rather than the family unit. For example, incarceration of the participating father is affecting him only as the participating mother continued her participation in the study.
Arm/Group | Intervention: Treatment as Usual + Focused Coparenting Consult | Control: Treatment as Usual
All-Cause Mortality (participants affected / at risk) | 3/140 | 1/136
Serious Adverse Events (participants affected / at risk) | 17/140 | 10/136
Other Adverse Events (participants affected / at risk) | 0/140 | 0/136
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention: Treatment as Usual + Focused Coparenting Consult (N=140) | Control: Treatment as Usual (N=136)
Incarceration (Social circumstances) | 7 (7) | 5 (5) — Participating mother is incarcerated for a short-term.
Death of Baby (Pregnancy, puerperium and perinatal conditions) | 3 (3) | 1 (1) — A child has passed away at birth or shortly after from birth/pregnancy complications. Children were not counted as participants in the study, only the parents were.
Domestic Violence (Social circumstances) | 3 (3) | 1 (1) — Participant father was incarcerated following a domestic violence episode against the participating mother.
DCF Removal of participating child (Social circumstances) | 0 (0) | 4 (4) — The participating child was removed by DCF.
Hospitalization (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — A child participant has been hospitalized due to respiratory issues and released home.
Baker Act (Psychiatric disorders) | 2 (2) | 0 (0) — A parent was hospitalized on a Baker Act (psychiatric hold) because of a suicidal ideation report to police.
Overdose (Psychiatric disorders) | 1 (1) | 0 (0) — Overdose by one of the participating parents.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (8):
  • Study Protocol (2020-07-06): https://cdn.clinicaltrials.gov/large-docs/91/NCT03097991/Prot_001.pdf
  • Statistical Analysis Plan (2022-01-31): https://cdn.clinicaltrials.gov/large-docs/91/NCT03097991/SAP_002.pdf
  • Informed Consent Form: Adult Consent Form (2020-03-27): https://cdn.clinicaltrials.gov/large-docs/91/NCT03097991/ICF_003.pdf
  • Informed Consent Form: Parental Consent Form (2020-03-27): https://cdn.clinicaltrials.gov/large-docs/91/NCT03097991/ICF_004.pdf
  • Informed Consent Form: Assent Form (2020-03-27): https://cdn.clinicaltrials.gov/large-docs/91/NCT03097991/ICF_005.pdf
  • Informed Consent Form: Adult Verbal Consent Form (2020-04-06): https://cdn.clinicaltrials.gov/large-docs/91/NCT03097991/ICF_006.pdf
  • Informed Consent Form: Verbal Parental Consent Form (2020-04-06): https://cdn.clinicaltrials.gov/large-docs/91/NCT03097991/ICF_007.pdf
  • Informed Consent Form: Verbal Assent Form (2020-04-06): https://cdn.clinicaltrials.gov/large-docs/91/NCT03097991/ICF_008.pdf